CLINICAL TRIAL: NCT00222898
Title: Pancreatic Cyst DNA Analysis
Brief Title: Cancer Detection in Pancreatic Cysts
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency); American Society for Gastrointestinal Endoscopy (Other)
Other Study IDs: PANDA
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2007-02

CONDITIONS: Pancreatic Cyst; Pancreatic Pseudocyst; Pancreatic Neoplasm
Keywords: Pancreatic Cyst; PANDA Study
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Pseudocyst; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: DNA analysis of pancreatic cyst fluid / buccal swab

SUMMARY:
The purpose of this study is to assist with early and accurate diagnosis of cancer in pancreatic cysts based on the analysis of DNA obtained by endoscopic ultrasound guided fine needle aspiration

DETAILED DESCRIPTION:
The study of pancreatic diseases is hindered by the organ's deep seated location and especially lack of symptoms during the early stages of disease development and progression e.g. pancreatic cancer. This is particularly true of pancreatic cysts, the variety and the malignant potential of which encompass a broad spectrum. The radiological features distinguishing a benign from a pre-malignant to a frankly malignant cyst in the pancreas are frequently underwhelming and have lead to the clinical practice of sampling all but the most obvious. The yield of the aspirate in turn is frequently not of a quality upon which a clinical decision can be based.

Most would agree that the best approach for management of pancreatic cystic neoplasm lies in early diagnosis, ideally at a precancerous stage. The effectiveness and applicability of this study is the based on the ability of the cyst DNA analysis to stratify the patients at risk of developing pancreatic cancer based on the extent of accumulated mutational damage.

ELIGIBILITY:
Inclusion Criteria:

* Previously scheduled for Endoscopic ULtrasound for evaluation of pancreatic cyst

Exclusion Criteria:

* Any condition that would preclude safe performance of EUS/FNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Asif Khalid, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (7):
  - Indiana University - Purdue University Indianapolis, Indianapolis, Indiana
  - Partners HealthCare System, Boston, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina